CLINICAL TRIAL: NCT01550484
Title: An Open Label, Multicenter Study, Evaluating the Safety and Efficacy of 18F-AV-133 PET Imaging to Identify Subjects With Dopaminergic Degeneration Among Subjects Presenting to a Movement Disorders Specialty Clinic With an Uncertain Diagnosis
Brief Title: A Trial of 18F-AV-133 Positron Emission Tomography (PET) Imaging to Differentiate Subjects With Parkinson's Disease (PD) From Other Movement Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-133-B04
Record Dates: First submitted 2012-03-06; First posted 2012-03-12 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Parkinson's Disease; Primary Parkinsonism; Lewy Body Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — florbenazine F 18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 18F-AV-133 — 222 MBq (6 mCi)

SUMMARY:
The purpose of this study is to determine whether 18F-AV-133 PET scans can be used to differentiate subjects with Parkinson's Disease from other movement disorders.

DETAILED DESCRIPTION:
The early detection and monitoring of neurodegenerative diseases including Parkinson's disease (PD), Alzheimer's disease (AD), Dementia with Lewy Bodies (DLB), and other dementias and movement disorders represent a very significant unmet medical need. Disease mechanisms are gradually becoming understood, and disease-modifying drugs are emerging that target the specific molecular pathology underlying each of these diseases. Tools for accurate and early differential diagnosis are thus necessary to determine the appropriate treatment for patients and to minimize inappropriate use of potentially harmful treatments. In addition, such diagnostic imaging tools are expected to permit monitoring of disease progression and will thus accelerate testing and development of disease-modifying drugs. Furthermore, the new imaging test may be useful as a prognostic tool by identifying humans suffering from neurodegenerative diseases before the clinical manifestations become evident.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 40 years of age;
* Presenting (within the last 3 months) for an initial evaluation to a movement disorders specialist with signs or symptoms suggestive of a movement disorder;
* The subject's signs or symptoms were previously evaluated by a physician who was not a movement disorders specialist during the previous six months;
* Absence of an established clinical movement disorder diagnosis;
* Symptoms mild in intensity, this includes Hoehn & Yahr ≤ 2 (Exceptions are allowed for subjects who meet criteria for Hoehn & Yahr stage 3 due to early onset of postural instability and/or gait impairment out of proportion to his/her other Parkinson signs and symptoms);
* Montreal Cognitive Assessment (MoCA) score ≥ 22;
* Can tolerate imaging visit procedures; and
* Provide written informed consent prior to study entry.

Exclusion Criteria:

* Have been referred to the movement disorders clinic primarily for the purpose of disease management (no diagnostic uncertainty exists on the part of the non-specialist or referring physician);
* Have a previous movement disorder diagnosis given by a movement disorders specialist prior to the time of enrollment;
* Have received a total of more than 90 days treatment with dopaminergic medications, including direct dopamine agonists or precursors (levodopa) or have received a total of more than 180 days treatment with MAO-B inhibitors, amantadine, anticholinergics or primidone or beta-blockers prescribed for treatment of tremor or signs of parkinsonism;
* Have had a sustained and clinically meaningful response to anti-parkinsonian medications;
* Are currently taking or have taken MAO-B inhibitors in the past 4 weeks;
* Have a known CNS structural lesion such as stroke or tumor that likely accounts for their symptoms;
* Have clinically meaningful cognitive impairment or dementia (mild cognitive problems as might be expected in the earliest stages of PD are not exclusionary);
* Have current clinically significant cardiovascular disease or clinically important abnormalities on screening ECG (including but not limited to QTc > 450 msec);
* Are currently taking medications that are known to cause QT-prolongation;
* Are currently taking medications with narrow therapeutic windows (e.g. warfarin or other anticoagulant therapies);
* Are currently taking tetrabenazine (TBZ), amphetamine type drugs;
* Have a current clinically significant endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer (excluding localized basal cell carcinoma and in situ prostate cancer) that would interfere with completion of the study;
* Have a recent history (within the past year) of alcohol or substance abuse or dependence;
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable contraception. Females must not be pregnant (negative serum beta-hCG at the time of screening and negative urine beta-hCG on the day of imaging), must not be breastfeeding at screening, must avoid becoming pregnant and use adequate contraceptive methods for 14 days prior to and 24 hours after administration of 18F-AV-133 for injection;
* Have had prior intracranial surgery; and
* Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of visual read of AV-133 PET scan vs. standard of truth | 18 months
  Sensitivity will be calculated as the percent of true positives which are correctly identified
  An expert, consensus diagnosis of PD performed by a panel of movement disorders specialists will be used as the standard of truth.
Specificity of visual read of AV-133 PET scan vs. standard of truth | 18 months
  Specificity will be calculated as the percent of true negatives which are correctly identified.
  An expert, consensus diagnosis of PD performed by a panel of movement disorders specialists will be used as the standard of truth.

SECONDARY OUTCOMES:
Inter-rater reliability of the visual read | 18 months
  Fleiss' kappa
Intra-rater reliability of the visual read | 18 months
  Intra-class kappa
Probability of progressive motor skill impairment | 18 months
  Compare rates of progressive impairment using PD rating scale in subjects with positive AV-133 PET scan vs. progressive impairment in subjects with negative AV-133 PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (15):
- United States (14):
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, New Haven, Connecticut
  - Research Site, Kansas City, Kansas
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Research Site, Sydney, New South Wales, Australia